CLINICAL TRIAL: NCT05923697
Title: The Feasibility and Potential Efficacy of Adding Addiction-focused EMDR to Regular Addiction Treatment A Multiple Baseline Study in Inpatients Who Use Non-opioid Drugs
Brief Title: Addiction-focused EMDR in Inpatients Who Use Non-opioid Drugs: a Multiple Baseline Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IrisZorg (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBS AF-EMDR NODD
Record Dates: First submitted 2023-06-13; First posted 2023-06-28 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
Keywords: Addiction; EMDR; Non-opioid drug disorder
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Study design: a non-concurrent multiple baseline design is used in which participants are allocated at random to a baseline period of 7, 10, or 13 days after which they proceed to an intervention phase of two weeks in which they receive four 90 min. sessions of AF-EMDR and a follow-up interview after one month. During both the baseline and the AF-EMDR intervention phase, participants also receive Treatment As Usual (TAU: Community Reinforcement Approach (CRA)), aimed at SUD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF-EMDR (Experimental): Intervention: a total of four 90 min. sessions of AF-EMDR twice per week added to TAU.
  Interventions: Behavioral: AF-EMDR

INTERVENTIONS:
Behavioral: AF-EMDR — Investigational treatment
  All participants receive four 90 min. AF-EMDR sessions within a timeframe of two weeks following the baseline phase. The AF-EMDR treatment will be provided by the principal investigators, a level II EMDR therapist (RvdH) and an EMDR consultant in training who developed the AF-EMDR protocol. The EMDR therapist (RvdH) will be trained by the EMDR consultant (WM), who is available for consultation. Additionally, both participate monthly in peer-supervision whereby videotaped sessions are discussed. See appendix 1 for a detailed understanding of the AF-EMDR protocol.

SUMMARY:
Rationale: It is well established that Substance Use Disorders (SUD) have severe health consequences. Despite behavioral and pharmacological treatment options, relapse rates remain high. In particular, for non-opioid drugs, such as amphetamines, cocaine, base-coke and cannabis, established, evidence-based pharmacological options to reduce craving, to substitute substance use or to enforce abstinence are lacking. Therefore, there is a need for effective interventions for patients who use non-opioid drugs to reach and maintain long-term abstinence.

A potential interesting intervention is addiction-focused Eye Movement Desensitization and Reprocessing (AF-EMDR) therapy. However, the limited research on AF-EMDR therapy and mixed findings thus far prohibit clinical use. Recently, on the basis of diverse findings thus far, an adjusted AF-EMDR therapy protocol has been developed.

DETAILED DESCRIPTION:
Objective: to investigate areas of uncertainty about a possible future pilot RCT using AF-EMDR as an add-on intervention in inpatients who use non-opioid drugs and receive regular, inpatient addiction treatment, by determining:

* Feasibility.
* Potential clinical efficacy.

Study population: adults with a primary non-opioid use disorder, who are admitted to an inpatient addiction care clinic. A total of nine eligible participants will be allocated (allocation ratio 1:1:1) at random, in a non-concurrent fashion to one of three baseline durations.

Intervention: a total of four 90 min. sessions of AF-EMDR twice per week added to TAU.

Main study parameters/endpoints:

* Feasibility issues.
* Changes in daily craving.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, patients must meet the following criteria:

Diagnosis of Tobacco Use Disorder according to the DSM-5 (American Psychiatric Association, 2013) criteria.

Age ≥ 18 years.

Good Dutch language proficiency (based on clinical judgement).

Smoking, on average, ≥ 10 cigarettes per day pre-admission.

A score of at least 5 on a scale from 0 to 10, for motivation and self-efficacy

A planned inpatient stay of ≥ 4 weeks.

Written informed consent.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

Serious therapy interfering behavior or symptoms that also interfere with TAU, based on clinical judgement (e. g. psychiatric or medical crisis that requires immediate intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants acceptability | 1 year
  The acceptability of AF-EMDR to participants in terms of compliance, measured by the total number of sessions attended and the proportion of attended versus non attended (planned) sessions; a higher proportion of attended sessions reflects better compliance.
Therapist acceptability | 1 year
  The acceptability of AF-EMDR to therapists in terms of adherence to the protocol, measured by the score of an independent rater on an a-priori established adherence rating protocol; a higher score reflects better adherence. Minimum=0 ;maximum=100
Study adherence of participants | 1 year
  from randomization until follow-up in terms of completion of tasks. A higher amount of completion means a better outcome.
Experienced (by participants) acceptability and burden | 1 year
  The number of experienced facilitators and barriers and subjective effectiveness of the AF-EMDR intervention.

SECONDARY OUTCOMES:
Change in: Subjective Units of Distress (SUD) | 1 year
  Within and/or over AF-EMDR sessions change in: Subjective Units of Distress (SUD) (Likert-type scales), a higher score reflects a worse outcome.
Change in craving | 1 year
  Within and/or over AF-EMDR sessions change in: Craving (Likert-type scale), a higher score reflects a worse outcome.
Change in Level of Urge (LoU) | 1 year
  Within and/or over AF-EMDR sessions change in: Change in Level of Urge (LoU), a higher score reflects a worse outcome.
Change in: Level of Positive Affect (LoPA) | 1 year
  Within and/or over AF-EMDR sessions change in: Level of Positive Affect (LoPA), a higher score reflects a better outcome.
changes in: Craving (MATE Q1: OCDS-5) | 1 year
  Baseline to follow-up assessment changes in: Craving (MATE Q1: OCDS-5), a higher score reflects a worse outcome
changes in: Craving-related self-control/self-efficacy (SCCQ) | 1 year
  Baseline to follow-up assessment changes in: Craving-related self-control/self-efficacy (SCCQ), a higher score reflects a worse outcome
changes in: Positive incentive value (SCCQ) | 1 year
  Baseline to follow-up assessment changes in: Positive incentive value (SCCQ), a higher score reflects a worse outcome
changes in: Substance use (past 30 days) (MATE section 1) | 1 year
  Baseline to follow-up assessment changes in: Substance use (past 30 days) (MATE section 1), a higher score reflects a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction clinic 'Tiel' IrisZorg, Tiel, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the final data collection and the journal in which these are published, we will decide on availability of IPD